CLINICAL TRIAL: NCT02343003
Title: A Prospective, Multi-Center, RCT Evaluating the Safety and Effectiveness of Coolief™ Cooled Radiofrequency Probe to Create Lesions of the Genicular Nerves and Comparing Corticosteroid Injection in the Management of Knee Pain
Brief Title: Nerve Ablation by Cooled Radiofrequency Compared to Corticosteroid Injection for Management of Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halyard Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105-14-0001
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2017-02

CONDITIONS: Osteoarthritis of the Knee
Keywords: cooled radiofrequency ablation; knee pain; osteoarthritis; pain management
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Agnosia | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cooled radiofrequency (Experimental): Cooled radiofrequency energy will be delivered to study subjects' knees to ablate culprit sensory nerves and reduce knee pain
  Interventions: Device: Cooled Radiofrequency
- Corticosteroid injection (Active Comparator): Corticosteroid injections will be administered to study subjects' knees to reduce knee pain
  Interventions: Drug: Corticosteroid injection

INTERVENTIONS:
Device: Cooled Radiofrequency — Delivery of energy to ablate sensory nerves via cooled radiofrequency probe
  Other Names: Coolief
  Arms: Cooled radiofrequency
Drug: Corticosteroid injection — Delivery of corticosteroid into knee by injection with needle to reduce knee pain
  Arms: Corticosteroid injection

SUMMARY:
This study is designed to:

* Determine the effectiveness (primarily measured by pain relief) of Coolief when used to create radiofrequency lesions of the genicular nerves compared to pain relief following corticosteroid injection; and
* Confirm the safety of Coolief when used to perform radiofrequency lesions of the genicular nerves in subjects to manage knee pain compared to safety of corticosteroid injection

DETAILED DESCRIPTION:
This is a prospective, randomized, multicenter comparison study examining the outcomes of subjects having knee pain undergoing a procedure to create a radiofrequency lesion of the genicular nerves with the Coolief system compared to subjects receiving corticosteroid injection. A total of approximately 144 subjects will be enrolled into this study with subjects undergoing either radiofrequency neurotomy or corticosteroid injection in a 1:1 randomization scheme. Follow up will be conducted for a total of 12 months post Coolief procedure with the primary endpoint being completed at month 6. Subjects randomized to the comparison (corticosteroid) group will have the option to cross over to the neurotomy group after completing the 6 month endpoint assessment. They would then be followed for an additional 6 months. Pain, overall outcome, quality of life, pain medication use, and adverse events will be compared between the two treatment groups in order to determine success.

Primary Effectiveness Endpoint:

The proportion of subjects whose knee pain is reduced by ≥ 50% based on the NRS scale at 6 Months.

Primary Safety Endpoint:

The proportion of subjects experiencing adverse events through final follow up.

Secondary Effectiveness Endpoints:

* The proportion of subjects whose knee pain is reduced from baseline by ≥ 50% based on the Numeric Rating Scale (NRS) at 12 months.
* Improvement in global outcome from baseline as measured by the Oxford Knee Score at 6 months and 12 months.

Tertiary Effectiveness Endpoint:

Subject satisfaction as measured by the Global Perceived Effect Score at 6 months and 12 months.

Quaternary Effectiveness Endpoint:

Reduction in pain medication usage from baseline as measured by subject self-reported average daily dosage.

In addition, exploratory analyses of health economic indicators may be performed.

Subjects will participate in the study for up to 13 months (2 week roll-in period + treatment visit + 12 month follow up), except for subjects who participate in the optional crossover group. These crossover subjects will be on study for up to 15 months (2 week roll-in + treatment + 6 month follow-up and crossover + 6 month follow up). Enrollment is anticipated to take approximately 6-8 months.

ELIGIBILITY:
INCLUSION CRITERIA

1. Age ≥ 21 years
2. Able to understand the informed consent form and provide written informed consent and able to complete outcome measures
3. History of chronic knee pain for longer than 6 months unresponsive to conservative treatments (PT, oral analgesics, intra-articular injections with steroids and/or viscosupplementation)
4. Positive response (defined as a decrease in numeric pain scores of at least 50%) to a geniculate nerve block of the index knee
5. Pain on NRS ≥ 6 on a 10 point scale for the index knee
6. Radiologic confirmation of osteoarthritis (x-ray/MRI/CT) of OA grade of 2 (mild), 3 (moderate) or 4 (severe) noted within 12 months for the index knee
7. Oxford Knee Score group at Baseline of ≤ 35 indicating moderate to severe OA in the index knee
8. If the patient is taking an opioid or other morphine equivalent medication, the dose must be considered clinically stable (defined as <10% change in dosage for ≥ 2 months prior to the screening visit).
9. Analgesics including membrane stabilizers such as Neurontin and antidepressants for pain such as Cymbalta must be clinically stable (defined as stable dosage for ≥ 6 weeks prior to the screening visit) and shall not change during the course of the study without approval of investigator. Agree to see one pain doctor (study investigator) for knee pain during the study period
10. Index knee pathology that is consistent with generally accepted indications for total knee arthroplasty.
11. Willing to delay any surgical intervention for the index knee for 12 months.
12. Willingness to provide informed consent and to comply with the requirements of this protocol for the full duration.

EXCLUSION CRITERIA

1. Pseudo arthritis, rheumatoid arthritis or other systemic inflammatory arthritis condition that could cause knee pain.
2. Previous or pending lower limb amputation.
3. Intra-articular steroid, platelet rich plasma (PRP) or hyaluronic acid injections in the index knee within 90 days from the screening visit.
4. An intra-articular corticosteroid injection is not indicated as an appropriate treatment option.
5. Prior radiofrequency of the genicular nerves of the index knee.
6. Prior partial, resurfacing, or total knee arthroplasty in index knee.
7. Clinically significant ligamentous laxity of the index knee.
8. Evidence of structural abnormality other than osteoarthritis of knee, hip or back that materially affects gait or function of the knee or is the underlying cause of the knee pain.
9. BMI > 40.
10. Extremely thin patients and those with minimal subcutaneous tissue thickness that would not accommodate a lesion of up to 14 mm in diameter to limit the risk of skin burns.
11. Pending or active compensation claim, litigation or disability remuneration (secondary gain) related to knee.
12. Pregnant or intent of becoming pregnant during the study period.
13. Chronic pain associated with significant psychosocial dysfunction.
14. Beck's Depression Index score of > 22 (indicates clinically depressed state).
15. Allergies to any of the medications to be used during the procedure.
16. Systemic or localized infection at needle entry sites (subject may be considered for inclusion once infection is resolved).
17. History of uncontrolled coagulopathy, ongoing coagulation treatment or unexplained or uncontrollable bleeding that is uncorrectable.
18. Identifiable anatomical variability that would materially alter the procedure as described in the protocol.
19. Within the preceding 2 years, subject has suffered from active narcotic addiction, substance or alcohol abuse.
20. Current prescribed opioid medications equivalent to greater than 60 morphine equivalent daily opioid dose.
21. Uncontrolled immunosuppression (e.g. AIDS, cancer, diabetes, etc.)
22. Subject currently implanted with pacemaker or defibrillator.
23. Participating in another clinical trial/investigation within 30 days prior to signing informed consent.
24. Subject unwilling or unable to comply with follow up schedule or protocol requirements.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David T Curd, MS, Study Director — Halyard Health, Inc.
Locations (11):
- United States (11):
  - Valley Anesthesiology Consultants - Estrella, Phoenix, Arizona
  - Valley Anesthesiology Consultants/Valley Pain Consultants, Scottsdale, Arizona
  - Orthopedic Pain Specialists, Santa Monica, California
  - Rush University Medical Center, Chicago, Illinois
  - MAPS Applied Research Center, Inc., Maple Grove, Minnesota
  - Ainsworth Institute of Pain Management, New York, New York
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Drexel University, Philadelphia, Pennsylvania
  - Piedmont Comprehensive Pain Management, Greenville, South Carolina
  - Virginia iSpine Physicians, Richmond, Virginia
  - Advanced Pain Management, Greenfield, Wisconsin

REFERENCES:
- [Derived] Davis T, Loudermilk E, DePalma M, Hunter C, Lindley DA, Patel N, Choi D, Soloman M, Gupta A, Desai M, Cook E, Kapural L. Twelve-month analgesia and rescue, by cooled radiofrequency ablation treatment of osteoarthritic knee pain: results from a prospective, multicenter, randomized, cross-over trial. Reg Anesth Pain Med. 2019 Feb 16:rapm-2018-100051. doi: 10.1136/rapm-2018-100051. Online ahead of print. PMID 30772821
- [Derived] Davis T, Loudermilk E, DePalma M, Hunter C, Lindley D, Patel N, Choi D, Soloman M, Gupta A, Desai M, Buvanendran A, Kapural L. Prospective, Multicenter, Randomized, Crossover Clinical Trial Comparing the Safety and Effectiveness of Cooled Radiofrequency Ablation With Corticosteroid Injection in the Management of Knee Pain From Osteoarthritis. Reg Anesth Pain Med. 2018 Jan;43(1):84-91. doi: 10.1097/AAP.0000000000000690. PMID 29095245

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cooled Radiofrequency | Corticosteroid Injection
Started | 76 | 75
Completed (Completion is with respect to the 6-month primary outcome.) | 58 | 68
Not Completed | 18 | 7
Not completed — Withdrawal by Subject | 9 | 4
Not completed — Lost to Follow-up | 5 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Death | 0 | 1
Not completed — exclusion criteria met | 1 | 1
Not completed — terminated by sponsor | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cooled Radiofrequency | Corticosteroid Injection | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 30 | 75
  >=65 years | 31 | 45 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (11.9) | 66.1 (13.1) | 64.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 49 | 99
  Male | 26 | 26 | 52
Region of Enrollment [Number; unit: participants]
  United States | 76 | 75 | 151

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS)
Description: The number of subjects whose knee pain is reduced by ≥ 50% based on the Numeric Rating Scale (NRS). The NRS is an 11-point scale (0 points to 10 points), where 0 points equals "no pain" and 10 points equals the "worst pain".
Time Frame: 6 months
Population: 58 of the 76 originally-randomized study subjects in the Cooled radiofrequency group completed this 6 month outcome. 68 of the originally-randomized 75 study subjects in the Corticosteroid injection group completed this 6 month outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency | Corticosteroid Injection
Number analyzed (Participants) | 58 | 68
Participants | 43 | 11

2. Primary Outcome: Safety: Number of Subjects Experiencing Adverse Events Through Final Follow up.
Description: Safety Endpoint: Number of subjects experiencing adverse events through final follow up.
Time Frame: 6 months and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency | Corticosteroid Injection
Number analyzed (Participants) | 76 | 75
Participants
  6 months post-intervention | 34 | 31
  12 months post-intervention | 12 | 3

3. Secondary Outcome: Numeric Rating Scale
Description: The number of subjects whose knee pain is reduced from baseline by ≥ 50% based on the Numeric Rating Scale (NRS) at 12 months. The NRS is an 11-point scale (0 points to 10 points), where 0 points equals "no pain" and 10 points equals the "worst pain".
Time Frame: 12 months
Population: 52 of the 76 originally-randomized study subjects in the Cooled radiofrequency group completed this 12 month outcome. 4 of the originally-randomized 75 study subjects in the Corticosteroid injection group completed this 12 month outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency | Corticosteroid Injection
Number analyzed (Participants) | 52 | 4
Participants | 34 | 2

4. Secondary Outcome: Oxford Knee Score
Description: Improvement in global outcome from baseline as measured by the Oxford Knee Score at 6 months and 12 months. The Oxford Knee Score is determined by a 12-question survey that measures knee function, and is scored on a scale that ranges from 0 - 48 points, with scores of 0 - 19 = "severe arthritis", 20 - 29 = "moderate to severe arthritis", 30 - 39 = "mild to moderate arthritis", and 40 - 48 = "satisfactory joint function".
Time Frame: 6 months and 12 months
Population: 58 of the 76 originally-randomized study subjects in the Cooled radiofrequency group completed this 6 month outcome. 67 of the originally-randomized 75 study subjects in the Corticosteroid injection group completed this 6 month outcome. 12 months: 52/76 in Cooled radiofrequency group and 3/75 in Corticosteroid injection group completed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cooled Radiofrequency | Corticosteroid Injection
Number analyzed (Participants) | 58 | 67
units on a scale
  6 months post-intervention | 18.5 (9.9) | 5.7 (8.9)
  12 months post-intervention: number analyzed (Participants) | 52 | 3
  12 months post-intervention | 17.3 (12) | 8.7 (9.9)

5. Other Pre Specified Outcome: Subject Satisfaction - Number of Participants With a Global Perceived Effect Score of 5 or Greater
Description: Subject satisfaction as measured by the Global Perceived Effect Score at 6 months and 12 months. The study subjects' perception of treatment effect was reflected by the Global Perceived Effect (GPE). The Global Perceived Effect is a 7-point scale: 1 point = "worst ever", 2 points = "much worse", 3 points = "worse", 4 points = "not improved but not worse", 5 points = "improved", 6 points = "much improved", 7 points = "best ever".
Time Frame: 6 months and 12 months
Population: 58 of the 76 originally-randomized study subjects in the Cooled radiofrequency group completed this 6 month outcome. 67 of the originally-randomized 75 study subjects in the Corticosteroid injection group completed this 6 month outcome. 12 months: 52/76 in Cooled radiofrequency group and 4/75 in Corticosteroid injection group completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cooled Radiofrequency | Corticosteroid Injection
Number analyzed (Participants) | 58 | 67
Participants
  6 months post-intervention | 53 | 16
  12 months post-intervention: number analyzed (Participants) | 52 | 4
  12 months post-intervention | 39 | 2

6. Other Pre Specified Outcome: Medication Usage
Description: Reduction in pain medication usage from baseline as measured by subject self-reported average daily dosage.
Time Frame: 6 months and 12 months
Population: 17 of the 76 originally-randomized study subjects in the Cooled radiofrequency group completed this 6 month outcome. 25 of the originally-randomized 75 study subjects in the Corticosteroid injection group completed this 6 month outcome. 12 months: 17/76 in Cooled radiofrequency group and 2/75 in Corticosteroid injection group completed.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Cooled Radiofrequency | Corticosteroid Injection
Number analyzed (Participants) | 17 | 25
milligrams
  6 months post-intervention | 2.4 (8.3) | -0.6 (9.8)
  12 months post-intervention: number analyzed (Participants) | 17 | 2
  12 months post-intervention | 1 (10.3) | 2.5 (17.7)

ADVERSE EVENTS:
Time Frame: 12 months
Description: A protocol-directed review of adverse events at pre-specified time points was conducted to collect the adverse events.
Arm/Group | Cooled Radiofrequency | Corticosteroid Injection
Serious Adverse Events (participants affected / at risk) | 3/76 | 9/75
Other Adverse Events (participants affected / at risk) | 43/76 | 25/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cooled Radiofrequency (N=76) | Corticosteroid Injection (N=75)
respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
urogenital (Renal and urinary disorders) | 1 (1) | 1 (1)
gastrointestinal (Gastrointestinal disorders) | 0 (0) | 3 (4)
other (General disorders) | 0 (0) | 2 (2) — Adverse events were monitored/assessed without regard to the specific adverse event term
procedure (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
infection (Infections and infestations) | 1 (1) | 0 (0)
cardiovascular (Cardiac disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cooled Radiofrequency (N=76) | Corticosteroid Injection (N=75)
extremities (General disorders) | 36 (46) | 18 (24) — infection, pain: treated knee, contralateral knee, both knees
blood/lymphatic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
endocrine/metabolic (Endocrine disorders) | 1 (1) | 1 (1)
gastrointestinal (Gastrointestinal disorders) | 3 (3) | 2 (5)
head, eyes, ears, nose, throat (General disorders) | 1 (1) | 2 (2)
musculoskeletal (Musculoskeletal and connective tissue disorders) | 8 (10) | 3 (5)
neurological (Nervous system disorders) | 2 (2) | 1 (3)
respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7)
skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
urogenital (Renal and urinary disorders) | 0 (0) | 2 (2)
other (General disorders) | 4 (6) | 6 (10) — Adverse events were monitored/assessed without regard to the specific adverse event term

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No